CLINICAL TRIAL: NCT03463304
Title: The Influence of Host Environmental Factors on the Gut Microbiome - Endocannabinoid Axis in Metabolic and Mental Health
Brief Title: Environmental Factors and the Gut Microbiome - Endocannabinoid Axis
Acronym: eMECA
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Alain Veilleux, Affiliated Professor, Laval University
Other Study IDs: 2017-328
Record Dates: First submitted 2018-02-20; First posted 2018-03-13 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Food Habits; Energy Metabolism; Mental Health Wellness 1; Intestinal Disease
Keywords: Gut Microbiota; endocannabinoide; Metabolic health; Gastrointestinal health; Mental wellbeing
MeSH Terms: conditions — Feeding Behavior; Intestinal Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal matter, blood and plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The general objective of this project is to investigate the interplay of the gut microbiome - endocannabinoid axis with host environmental factors and intestinal, metabolic and mental health status in free-living adults with various metabolic statuses and lifestyles.

DETAILED DESCRIPTION:
The gut microbiome and the endocannabinoid system (ECS) could be interacting together and influence local enteric and peripheral metabolic functions and mental health.

The association of some host environmental factors (e.g. age, metabolic status, dietary habits) with gut microbiota composition and function has been investigated but, to our knowledge, little is known about their influence on the ECS.

There is also a need to better understand the influence of these factors and the interplay between the gut microbiota and the ECS and their relationship with intestinal, metabolic and mental health.

The investigators therefore propose to fill this knowledge-gap in the general population of adults with various body composition, dietary habits and daily physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* Computer and internet access
* Understanding of written French

Exclusion Criteria:

* Intestinal pathologies
* Pregnancy or breast-feeding
* Recent significant weight variations
* Recent completion of antibiotic treatment
* Alcohol consumption over sex-specific recommendations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Free-living adults with various body composition, dietary habits and daily physical activity levels from the Quebec city region.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the influence of dietary habits assessed via Food Frequency Questionnaire (FFQ) on the relationship between gut microbiota composition and circulating endocannabinoids | September 2018
  FFQ items will be used to identify dietary habits by unsupervised clustering to evaluate their association with gut microbiota composition obtained from ribosomal RNA sequencing and plasma endocannabinoid (e.g. Arachidonoylethanolamide, 2 arachidonoyl glycerol and their derivatives) concentrations.

SECONDARY OUTCOMES:
Evaluation of the effect of adiposity assessed by Dual-energy X-ray Absorptiometry (DXA) scan on the relationship between gut microbiota composition and circulating endocannabinoids. | September 2018
  The effect of adiposity measured by DXA scan on the relationship between gut microbiota composition and diversity obtained from ribosomal RNA sequencing and plasma endocannabinoids (e.g. Arachidonoylethanolamide, 2 arachidonoyl glycerol and their derivatives) will be investigated.
Evaluation of the effect of fasting glycemia on the relationship between gut microbiota composition and circulating endocannabinoids. | September 2018
  The effect of fasting glycemia, used to infer metabolic status, on the relationship between gut microbiota composition and diversity obtained from ribosomal RNA sequencing and plasma endocannabinoids (e.g. Arachidonoylethanolamide, 2 arachidonoyl glycerol and their derivatives) will be investigated.
Evaluation of the effect of fasting triglyceridemia on the relationship between gut microbiota composition and circulating endocannabinoids. | September 2018
  The effect of fasting triglyceridemia, used to infer metabolic status, on the relationship between gut microbiota composition and diversity obtained from ribosomal RNA sequencing and plasma endocannabinoids (e.g. Arachidonoylethanolamide, 2 arachidonoyl glycerol and their derivatives) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Veilleux, PhD, Principal Investigator — Laval University
Locations (1):
- Institut sur la nutrition et les aliments fonctionnels - INAF, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided